CLINICAL TRIAL: NCT04527770
Title: Midazolam Versus Dexamethasone as an Adjuvant to Local Anesthetics in the Ultrasound Guided Hydrodissection of Median Nerve for Treatment of Carpal Tunnel Syndrome Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mina Maher, Principle investigator, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 644/4-2020
Record Dates: First submitted 2020-08-23; First posted 2020-08-27 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Pain Syndrome
Keywords: Midazolam; median nerve; dexamethasone
MeSH Terms: conditions — Somatoform Disorders | interventions — Dexamethasone; Midazolam

STUDY DESIGN:
Intervention Model Description: 2 groups received hydrodissection sonar guided , one group received 50 mic/kg midazolam and the other received 8 mg dexamethasone
Who Masked: Participant, Investigator
Masking Description: both drugs are the same colour and volume injected by a staff member not aware of study design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dexamethasone group (Active Comparator): sonar guided median nerve hydrodissection by bupivacaine 0.5% and dexamethasone
  Interventions: Drug: Dexamethasone
- midazolam group (Active Comparator): sonar guided median nerve hydrodissection by bupivacaine 0.5% and midazolam
  Interventions: Drug: Midazolam injection

INTERVENTIONS:
Drug: Dexamethasone — Ultrasound guided median nerve hydrodiseection using dexamethasone or midazolam
  Other Names: midazolam
  Arms: dexamethasone group
Drug: Midazolam injection — intracarpal injection of midazolam and bupivacaine 0.5%
  Arms: midazolam group

SUMMARY:
midazolam and dexamethasone both can counteract chronic pain. either via GABA mimetic action or via anti prostaglandins

DETAILED DESCRIPTION:
Entrapement syndrome - namely median nerve compression in carpal tunnel syndrome - causes chronic pain that can be refractory to medical treatment . Ultrasound guided hydrodissection is an option for alleviating pain . Recurrence is the main side effect of injection. We try in this research to prevent recurrence rate . Midazolam and dexamethasone both are used in chronic pain . Midazolm act by GABA mimetic action while dexamethasone act by decrease interleukin formation

ELIGIBILITY:
Inclusion Criteria:

* numbness or pain in the nerve distribution, nerve conduction studies (NCS) corresponding with AANEM guidelines
* Nerve cross sectional area >12mm2

Exclusion Criteria:

* Refusal to participate
* History of operation in median nerve.were patient refusal to participate, pain recurrence after previous injection and severe symptoms requiring surgical release, diabetic patients

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
comparing efficacy of midazolam against dexmethasone in combination with bupivacaine 0.5% | up to 6 months
  use of visual analogue score

SECONDARY OUTCOMES:
Subjective pain assesment | up to 6 months
  BOSTON questionnaire
complications | pain recurrence after 6 months, neurotoxicity immediately after injection
  neurotoxicity, pain recurrence after injection
Nerve electrophysiology | up to 6 months
  sensory nerve conduction , distal motor latency.
nerve sonogram | up to 6 months
  nerve cross sectional area.

CONTACTS AND LOCATIONS:
Locations (1):
- Mina Maher Raouf, ALMinya, Egypt, Egypt